CLINICAL TRIAL: NCT00559858
Title: A Randomised Placebo-controlled Study Evaluating the Role of Pyridoxine in Controlling Capecitabine-induced Hand-foot Syndrome
Brief Title: Pyridoxine in Preventing Hand-Foot Syndrome in Patients Who Are Receiving Capecitabine for Advanced Colorectal Cancer or Breast Cancer
Status: Unknown | Phase: Phase 3 | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: Cambridge University Hospitals NHS Foundation Trust (Other)
Organization: National Cancer Institute (NCI) (NIH)
Allocation: Randomized | Masking: Double | Purpose: Supportive Care
Other Study IDs: CRCA-CCTC-CAPP-IT; CDR0000576453 (Registry Identifier: PDQ (Physician Data Query)); EUDRACT-2004-000325-29; EU-20786; ISRCTN82842634; CCLG-CAPP-IT
Record Dates: First submitted 2007-11-15; First posted 2007-11-16 (Estimated); Last update posted 2013-08-02 (Estimated); Status verified 2008-12

CONDITIONS: Breast Cancer; Colorectal Cancer; Palmar-plantar Erythrodysesthesia
Keywords: palmar-plantar erythrodysesthesia; breast cancer; male breast cancer; colon cancer; rectal cancer
MeSH Terms: conditions — Breast Neoplasms; Colorectal Neoplasms; Hand-Foot Syndrome; Breast Neoplasms, Male; Colonic Neoplasms; Rectal Neoplasms | interventions — Pyridoxine

INTERVENTIONS:
Dietary Supplement: pyridoxine hydrochloride
Other: placebo
Procedure: quality-of-life assessment

SUMMARY:
RATIONALE: Pyridoxine (vitamin B6) may prevent or lessen hand-foot syndrome caused by chemotherapy. It is not yet known whether pyridoxine is more effective than a placebo in preventing hand-foot syndrome.

PURPOSE: This phase III randomized trial is studying pyridoxine to see how well it works compared to a placebo in preventing hand-foot syndrome in patients who are receiving capecitabine for advanced colorectal cancer or breast cancer.

DETAILED DESCRIPTION:
OBJECTIVES:

Primary

* Determine whether pyridoxine can reduce the incidence of capecitabine dose modifications (dose delay and dose reductions) due to toxicity.

Secondary

* Determine the incidence of hand-foot syndrome (HFS).
* Determine the overall toxicity.
* Determine the quality of life.
* Determine the response to chemotherapy.
* Determine the progression-free survival.
* Determine the level of biomarkers which might predict the occurrence of HFS.

OUTLINE: This is a multicenter study. Patients are stratified according to disease (breast cancer vs colorectal cancer). Patients are randomized to 1 of 2 treatment arms.

* Arm I: Patients receive oral pyridoxine hydrochloride 3 times daily beginning with the initiation of capecitabine chemotherapy and continuing until completion of chemotherapy.
* Arm II: Patients receive oral placebo 3 times daily beginning with the initiation of capecitabine chemotherapy and continuing until completion of chemotherapy.

In both arms, treatment continues in the absence of disease progression or unacceptable toxicity.

Evidence of hand-foot syndrome is assessed at baseline and before each course of capecitabine. Quality of life is assessed at baseline and then every 6 weeks.

After completion of study treatment, patients are followed at 6 and 12 weeks.

ELIGIBILITY:
DISEASE CHARACTERISTICS:

* Diagnosis of advanced colorectal or breast carcinoma

  * Hormone receptor status not specified
* Receiving single-agent capecitabine chemotherapy
* Measurable disease for response assessment, determined on an individual patient basis, using conventional clinical and/or radiological methods

PATIENT CHARACTERISTICS:

* ECOG performance status 0-2
* Menopausal status not specified
* Life expectancy ≥ 12 weeks
* Hemoglobin ≥ 10 g/dL
* Platelet count ≥ 100,000 mm^3
* WBC ≥ 3,000/mm^3
* ANC ≥ 1,500/mm^3
* Bilirubin ≤ 1.3 x upper limit of normal (ULN)
* Alkaline phosphatase ≤ 5 x ULN
* AST and ALT ≤ 5 x ULN
* Creatinine ≤ 1.5 x ULN
* Not pregnant or nursing
* Negative pregnancy test
* Fertile patients must use effective contraception during and for 3 months after completion of study treatment
* No other serious or uncontrolled illness which, in the opinion of the investigator, makes it undesirable for the patient to enter the trial
* No medical or psychiatric condition which would influence the ability to provide informed consent

PRIOR CONCURRENT THERAPY:

* See Disease Characteristics
* At least 6 weeks since prior investigational agents
* Concurrent radiotherapy allowed
* No other concurrent chemotherapy or immunotherapy
* No concurrent nonsteroidal anti-inflammatory drugs NSAIDs) for the primary purpose of treating hand-foot syndrome (HFS) or cancer

  * NSAIDs for conditions other than HFS or cancer allowed

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2004-12; Primary Completion 2009-12 (Estimated)

PRIMARY OUTCOMES:
Incidence of capecitabine dose modifications (dose delay and dose reductions) due to toxicity

SECONDARY OUTCOMES:
Incidence of hand-foot syndrome (HFS)
Overall toxicity
Quality of life
Response to chemotherapy
Progression-free survival
Measurement of biomarkers that might predict the occurrence of HFS

CONTACTS AND LOCATIONS:
Overall Officials: Pippa Corrie, PhD, FRCP, Study Chair — Cambridge University Hospitals NHS Foundation Trust
Locations (16):
- United Kingdom (16):
  - Basildon University Hospital, Basildon, England
  - Primrose Oncology Unit, Bedford, England
  - West Suffolk Hospital, Bury St Edmunds, England
  - Addenbrooke's Hospital, Cambridge, England
  - Kent and Canterbury Hospital, Canterbury, England
  - Derbyshire Royal Infirmary, Derby, England
  - Royal Devon and Exeter Hospital, Exeter, England
  - Queen Elizabeth Hospital, Kings Lynn, England
  - Royal Albert Edward Infirmary, Lancanshire, England
  - Mid Kent Oncology Centre at Maidstone Hospital, Maidstone, England
  - Peterborough Hospitals Trust, Peterborough, England
  - Derriford Hospital, Plymouth, England
  - Kent and Sussex Hospital, Royal Tunbridge Wells, England
  - Great Western Hospital, Swindon, England
  - Walsall Manor Hospital, Walsall, England
  - Southend University Hospital NHS Foundation Trust, Westcliff-on-Sea, England